CLINICAL TRIAL: NCT07148765
Title: The Feasibility of Using Wearable Electronic Devices Following Cystectomy to Identify Early Biometric Signatures of Readmission
Brief Title: Use of Wearables Following Cystectomy- Part II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Epstein, Fellow, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25060009
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Neurogenic Bladder Disorder; Cystectomy
Keywords: Wearable Electronic Devices; Patient Reported Outcome Measures; Postoperative Care; Remote Monitoring; Cystectomy; Urinary Diversion; Fitbit
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fitbit Sense 2 + smartphone surveys (Experimental): Participants undergoing remote monitoring following cystectomy using Fitbit sense 2 device for continuous biometric marker collection and transmission and completion of daily PRO questionnaires administered via smartphone application to trigger provider response within 24 hours of predefined threshold abnormalities.
  Interventions: Device: Fitbit Sense 2; Other: Smartphone application survey

INTERVENTIONS:
Device: Fitbit Sense 2 — Continuous biometric monitoring (e.g., heart rate, pulse oximetry, respiratory rate, etc.) that will trigger alerts based on predefined threshold criteria for health care providers to respond to by contacting patients within 24 hours of alert.
Other: Smartphone application survey — Daily questionnaire to record PROs will be administered via patient smartphones. Concerning PROs will trigger alerts which health care providers will respond to by contacting patients within 24 hours of alert.

SUMMARY:
The goal of this observational study is to learn about the practical considerations for having health care providers respond in real-time to abnormalities detected remotely for patients recovering from cystectomy following discharge from the hospital. Participants will be asked to wear a wearable fitness tracker (e.g., Fitbit) and answer a daily brief questionnaire on their smartphone.

The main question[s] the investigators aims to answer are:

* Is it practical to have health care providers respond in real-time to abnormal biomarkers collected using fitness trackers for patients recovering from cystectomy?
* Can we identify early biomarker signatures (e.g. using heart rate, pulse oximetry, respiratory rate, etc.) that can predict adverse events that lead to hospital readmissions?

Participants will

* Set up and use a Fitbit Sense 2 device for up to 2 weeks prior to surgery and again for 30 days following discharge after their surgical hospitalization.
* Download and complete questionnaires in a smartphone application for up to 2 weeks prior to surgery and again for 30 days following discharge after their surgical hospitalization.
* Trigger automated alerts when abnormal biometric data (from the Fitbit device) or concerning survey responses are detected.
* Receive contact from a health care provider within 24 hours of an automated alert being generated.

DETAILED DESCRIPTION:
Cystectomy is associated with high rates of complications and readmissions, with approximately one-quarter of patients readmitted within 30 days. Despite advances in perioperative care, these rates have remained unchanged. Remote patient monitoring using a combination of consumer-grade wearable electronic devices, such as the Fitbit Sense 2, and smartphone application administered questionnaires offers an accessible method for continuous, passive collection of digital biomarkers (e.g., heart rate, respiratory rate, SpO2, step count, sleep patterns) and collection of patient-reported outcomes (PROs) in the outpatient setting. Prior studies have demonstrated the feasibility of wearable devices and electronic PRO monitoring postoperatively, but limited data exist on the real-time use of biomarker and PRO data to trigger provider responses in cystectomy patients following discharge.

The investigators' primary objective is to evaluate the feasibility of investigating continuous remote monitoring using wearable electronic devices and smartphone application-administered questionnaires to trigger real-time alerts to abnormalities in digital biomarkers and PROs in the 30-day postoperative period following cystectomy. The secondary objective of this study is to identify early biometric signatures predictive of adverse events that lead to readmissions.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Owns a smartphone
* Scheduled to undergo cystectomy with urinary diversion at a UPMC hospital

Exclusion Criteria:

* No reliable internet access
* Concurrent enrollment in another interventional study that may interfere with outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who remain in the study from enrollment until trial completion (participant retention) | From enrollment to 30 days post-discharge following cystectomy hospitalization
Participant wearable electronic device adherence | From day of discharge following cystectomy hospitalization to 30 days post-discharge
  Proportion of patients who wear and transmit data from the provided Fitbit Sense 2 device for at least 16 hours per day for more 14 days

SECONDARY OUTCOMES:
Number of participants readmitted | from discharge following cystectomy hospitalization to 30-days post-discharge
Number of participant unplanned encounters | From time of discharge following cystectomy hospitalization to 30 days post-discharge
  Any unscheduled interaction with healthcare provider triggered by either the patient or a healthcare provider, including initiated by study alerts. This includes emergency department visits, telemedicine visits, telephone encounters, urgent care visits, unscheduled outpatient clinic visits, and hospital readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Epstein, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: The data will be available at the time of publication and 7 years following (as data stored at institution for 7 years following project completion).
Access Criteria: Interested researcher can contact the study team for any purpose. Individual participant data to researchers who provide a methodologically sound proposal. The data will be made available following a data use agreement.